CLINICAL TRIAL: NCT02731716
Title: Transforming Primary Care Payment in Hawaii
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Hawaii Medical Service Association (Other)
Responsible Party: Principal Investigator, Amol Navathe, MD, PHD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 823981
Record Dates: First submitted 2016-03-28; First posted 2016-04-07 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- New Payment Model (Experimental): Providers in the first arm will no longer be paid based upon FFS, but on the new payment model. Providers will receive a PMPM payment for attributed members, a quality incentive payment based upon attainment of sixteen quality metrics, and a possible bonus payment for savings in total cost of care at the provider organization level.
  Interventions: Behavioral: New Payment Model
- Social Comparisons (Experimental): Providers will no longer be paid based upon FFS, but on the new payment model. Providers will receive a PMPM payment for attributed members, a quality incentive payment based upon attainment of sixteen quality metrics, and a possible bonus payment for savings in total cost of care at the provider organization level. Providers will also receive weekly emails that will show comparisons of their own performance against their peers within the same provider organization on specific quality measures and total cost of care.
  Interventions: Behavioral: New Payment Model; Behavioral: Social Comparisons
- A1c Member/Provider Incentive (Experimental): Providers will no longer be paid based upon FFS, but on the new payment model, which includes a PMPM payment for attributed members, a quality incentive payment based upon attainment of quality metrics, and a possible bonus payment for savings in total cost of care. Providers will also receive weekly emails that will show comparisons of their own performance against their peers within the same provider organization on specific quality measures and total cost of care. There is also a shared incentive between the member and the provider. The member incentive will be a payment made to diabetic patients with an A1C of greater than or equal to 9% who experience a reduction of at least 0.5%. Each participating member and PCP can receive up to $75 per quarter for A1C reduction.
  Interventions: Behavioral: New Payment Model; Behavioral: Social Comparisons; Behavioral: A1c Member/Provider Incentive

INTERVENTIONS:
Behavioral: New Payment Model — Providers will no longer be paid based upon FFS, but on the new payment model, which includes PMPM and quality incentives.
Behavioral: Social Comparisons — Providers will receive weekly emails showing comparisons in quality metrics and total cost of care. They will be compared to other providers in their provider organization.
  Arms: A1c Member/Provider Incentive; Social Comparisons
Behavioral: A1c Member/Provider Incentive — Attributed members and their PCPs will receive up to $75 for a reduction of a1c by 0.5% per quarter (2 quarters).
  Arms: A1c Member/Provider Incentive

SUMMARY:
To design an innovative payment system that improves upon fee-for-service (FFS), incorporates behavioral economic principles, and improves work satisfaction among primary care physicians (PCPs) while improving quality and reducing health spending at the state level. Second, to test the incremental effectiveness of two additional interventions: (1) shared financial incentives between physicians and poorly controlled diabetes and (2) social comparisons ranking physicians on quality metric performance and total cost of care.

DETAILED DESCRIPTION:
The goal of this project is to transform the Hawaii Medical Service Association (HMSA) primary care provider payment model to better incentive population health while bending the increasing trend of health spending in the state. Primary care and overall spending patterns will be studied to lay the foundation for a more rationally designed model. This model deliberately shifts away from FFS and includes three components: 1) a risk-adjusted per-member, per-month (PMPM) base payment, 2) an enhanced quality incentive program with larger bonus amounts and 3) a total cost of care incentive at the PO level. The aim is to build on the success of the Alternative Quality Contract (AQC) program implemented by Blue Cross Blue Shield (BCBS) of Massachusetts. While the AQC is used as a starting point, the study introduces and tests a number of innovations using concepts from behavioral economics. First, the move away from the FFS chassis to a PMPM-based capitated payment. Second, 20% of the PMPM payment is at-risk based on metrics designed to increase engagement between HMSA and physicians and engagement with performance feedback. Third, the number of metrics in the quality incentive program is drastically reduced from over 60 metrics to 10-12 per specialty. Fourth, the scoring of quality incentives incorporates rewards for improvement, rather than exclusively attainment of thresholds, to activate physicians along the entire performance distribution. In addition to implementing the new payment model, the initial experiment will include a test of two additional behavioral concepts: social comparisons for physicians and a shared incentive for physicians and poorly controlled diabetics tied to improve glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* HMSA physicians who are part of a Provider Organization that is participating in the payment transformation pilot.

Exclusion Criteria:

* Any physician who is not part of a participating Provider Organization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in Provider Performance | 1 year
  Provider performance on quality metrics will be compared across all three arms.

SECONDARY OUTCOMES:
Improvement in A1C among poorly controlled diabetics | 6 Months
  A1c levels will be compared across all three arms to see if there is a reduction in a1c in arm 3.
Primary Care Spending | 1 year
  Primary care spending in primary care providers will be compared across all three arms.

IPD SHARING:
Plan to Share IPD: No